CLINICAL TRIAL: NCT00500071
Title: A Prospective, Open-Label, Multi-Center, Dose-Optimization Study Evaluating the Efficacy, Safety and Tolerability of Vyvanse (Lisdexamfetamine Dimesylate) 20-70mg in Children Aged 6-12 Diagnosed With ADHD
Brief Title: Dose-Optimization Study Evaluating the Efficacy, Safety and Tolerability of Vyvanse (Lisdexamfetamine Dimesylate) in Children Aged 6-12 Diagnosed With ADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD489-310
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Results first posted 2009-09-01 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Vyvanse (lisdexamfetamine dimesylate)

INTERVENTIONS:
Drug: Vyvanse (lisdexamfetamine dimesylate) — Vyvanse™ 20mg once daily at 7 a.m.; dose increased weekly by 10mg until an acceptable response is achieved. Titration may proceed to a maximum daily dose 70mg/day.

SUMMARY:
Assess the efficacy & tolerability of Vyvanse when children aged 6-12 years diagnosed with ADHD are dosed to optimal effect.

DETAILED DESCRIPTION:
Dose-Optimization Study Evaluating the Efficacy, Safety and Tolerability of Vyvanse (lisdexamfetamine dimesylate) in Children aged 6-12 Diagnosed with ADHD

ELIGIBILITY:
Inclusion Criteria

1. Subject is a male or female aged 6-12 years inclusive at the time of consent.
2. Females of Child-bearing Potential (FOCP) must have a negative serum beta Human Chorionic Gonadotropin (HCG) pregnancy test at Screening and a negative urine pregnancy test at Baseline and agree to comply with any applicable contraceptive requirements of the protocol.
3. primary diagnosis of ADHD based on a detailed psychiatric evaluation.
4. Subjects must have a baseline ADHD-RS-IV total score ≥28.
5. Subject is functioning at an age-appropriate level intellectually.
6. comply with all the testing and requirements.
7. Subject is able to swallow a capsule.
8. Subject has blood pressure measurements within the 95th percentile for age, gender, and height.

Exclusion Criteria

1. Subject has a current, controlled (requiring a restricted medication) or uncontrolled, comorbid psychiatric diagnosis with significant symptoms such as Post Traumatic Stress Disorder, psychosis, bipolar illness, pervasive developmental disorder, severe obsessive compulsive disorder, severe depressive or severe anxiety disorder or other symptomatic manifestations.
2. Subject has Conduct Disorder.
3. Subject has a documented allergy, hypersensitivity, or intolerance to amphetamines.
4. Subject has failed to respond to one or more adequate courses (dose and duration) of amphetamine therapy.
5. The subject has a recent history (within the past 6 months) of suspected substance abuse or dependence.
6. Subject has a positive urine drug result.
7. Subject weighs less than 50 pounds (22.7kg).
8. Subject is significantly overweight.
9. Subject has a history of seizures (exclusive of febrile seizures), a tic disorder, a current diagnosis and/or family history of Tourette's Disorder.
10. Subject has any reported history of abnormal thyroid function.
11. Subject has taken another investigational product or taken part in a clinical trial within 30 days prior to Screening.
12. Subject has a concurrent chronic or acute illness (such as severe allergic rhinitis or an infectious process requiring antibiotics), disability, or other condition that might confound the results of safety assessments.
13. The female subject is pregnant or lactating.
14. Subject is well-controlled on their current ADHD medication with acceptable tolerability.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 318 (Actual)
Dates: Start 2007-06-28 (Actual); Primary Completion 2008-01-02 (Actual); Study Completion 2008-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (46):
- United States (46):
  - Melmed Center, Scottsdale, Arizona
  - Valley Clinical Research, El Centro, California
  - Peninsula Research Assoc, Inc, Rolling Hills Estates, California
  - UCSF-Langely Porter Psych Institute, San Francisco, California
  - Encompass Clinical Research, Spring Valley, California
  - Shire Clinical Research Site, Wildomar, California
  - Sarkis Clinical Trials, Gainesville, Florida
  - Shire Clinical Research Site, Hialeah, Florida
  - CNS Research Institute, Inc, Jacksonville, Florida
  - CORE Research, Inc, Maitland, Florida
  - Miami Research Associates, Miami, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Janus Center for Psychiatric Research, West Palm Beach, Florida
  - Children's Development Center, Winter Park, Florida
  - Capstone Clinical Research, Libertyville, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Shire Clinical Research Site, Terre Haute, Indiana
  - Shire Clinical Research Site, Newton, Kansas
  - Psychiatric Associates, Overland Park, Kansas
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Shire Clinical Research Site, Lexington, Kentucky
  - Pedia Research, Owensboro, Kentucky
  - Four Rivers Clinical Research, Inc., Paducah, Kentucky
  - Shire Clinical Research Site, Troy, Michigan
  - University of Rochester, School of Medicine and Dentistry, Rochester, New York
  - Piedmont Neuropsychiatry, Charlotte, North Carolina
  - University Commons Office Park, Durham, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - BHI, Inc., Moore, Oklahoma
  - Shire Clinical Research Site, Oklahoma City, Oklahoma
  - Oregon Center for Clinical Investigations, Inc, Eugene, Oregon
  - Oregon Center For Clinical Investigations, Inc., Portland, Oregon
  - Summit Research Network, Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc., Salem, Oregon
  - ADHD Program, Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania
  - The Jackson Clinic, Jackson, Tennessee
  - Clinical Neuroscience Solutions, Inc, Memphis, Tennessee
  - FutureSearch Trials, Austin, Texas
  - Claghorn-Lesem Research Clinic Inc., Bellaire, Texas
  - Red Oak Psychiatry Associates P.A., Houston, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - ADHD Clinic of San Antonio, San Antonio, Texas
  - NeuroScience, Inc, Herndon, Virginia
  - Dominion Clinical Research, Midlothian, Virginia
  - International Clinical Research Associates, LLC, Richmond, Virginia
  - Eastside Therapeutic Resource, Kirkland, Washington

REFERENCES:
- [Result] Findling RL, Ginsberg LD, Jain R, Gao J. Effectiveness, safety, and tolerability of lisdexamfetamine dimesylate in children with attention-deficit/hyperactivity disorder: an open-label, dose-optimization study. J Child Adolesc Psychopharmacol. 2009 Dec;19(6):649-62. doi: 10.1089/cap.2008.0165. PMID 20035583
- [Result] Katic A, Ginsberg L, Jain R, Adeyi B, Dirks B, Babcock T, Scheckner B, Richards C, Lasser R, Turgay A, Findling RL. Clinically relevant changes in emotional expression in children with ADHD treated with lisdexamfetamine dimesylate. J Atten Disord. 2012 Jul;16(5):384-97. doi: 10.1177/1087054710389990. Epub 2010 Dec 20. PMID 21173426
- [Result] Turgay A, Ginsberg L, Sarkis E, Jain R, Adeyi B, Gao J, Dirks B, Babcock T, Scheckner B, Richards C, Lasser R, Findling RL. Executive function deficits in children with attention-deficit/hyperactivity disorder and improvement with lisdexamfetamine dimesylate in an open-label study. J Child Adolesc Psychopharmacol. 2010 Dec;20(6):503-11. doi: 10.1089/cap.2009.0110. PMID 21186969
- See also: FDA recall information — http://www.fda.gov/opacom/7alerts.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study had three phases; 1)screening and wash-out; 2) dose-optimization (5 weeks) and maintenance (2 weeks); 3) 30-day safety follow-up. Dosing ranged from 20-70 mg once daily of Vyvanse.
Groups:
- Vyvanse: Lisdexamfetamine dimesylate (LDX)
Period: Screening and Washout Phase
Arm/Group | Vyvanse
Started | 318
Completed | 317
Not Completed | 1
Not completed — Protocol Violation | 1
Period: Dose-optimization and Maintenance Phase
Arm/Group | Vyvanse
Started | 317 (Safety population (i.e., received at least one dose of study medication))
Completed | 295
Not Completed | 22
Not completed — Adverse Event | 13
Not completed — Protocol Violation | 2
Not completed — Lack of Efficacy | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lack of protocol compliance | 4
Period: 30-day Safety Follow-up
Arm/Group | Vyvanse
Started | 295
Completed | 278
Not Completed | 17
Not completed — Lost to Follow-up | 17

BASELINE CHARACTERISTICS:
Arm/Group | Vyvanse
Number analyzed (Participants) | 318
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 318
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.1 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 225
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 318

OUTCOME MEASURES:

1. Secondary Outcome: Weekly Change From Baseline in Total ADHD-RS-IV Score
Description: Change in the Attention Deficit Hyperactivity Disorder Rating Scale-fourth edition (ADHD-RS-IV) total score from baseline. The ADHD-RS-IV consists of 18 items scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms) with total score ranging from 0 to 54.
Time Frame: Baseline and 1, 2, 3, 4, 5, 6, and 7 weeks
Population: ITT
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Vyvanse
Number analyzed (Participants) | 316
Units on a scale
  Week 1 | -11.3 (0.62)
  Week 2 | -17.8 (0.63)
  Week 3 | -21.7 (0.61)
  Week 4 | -25.4 (0.61)
  Week 5 | -27.0 (0.60)
  Week 6 | -28.9 (0.60)
  Week 7 | -29.8 (0.58)
Statistical Analysis 1: Comparison: Vyvanse; Week 1; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided
Statistical Analysis 2: Comparison: Vyvanse; Week 2; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided
Statistical Analysis 3: Comparison: Vyvanse; Week 3; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided
Statistical Analysis 4: Comparison: Vyvanse; Week 4; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided
Statistical Analysis 5: Comparison: Vyvanse; Week 5; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided
Statistical Analysis 6: Comparison: Vyvanse; Week 6; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided
Statistical Analysis 7: Comparison: Vyvanse; Week 7; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided

2. Primary Outcome: Change From Baseline in Total Attention Deficit Hyperactivity Disorder Rating Scale-fourth Edition (ADHD-RS-IV) Score at 7 Weeks
Description: as for outcome 1
Time Frame: Baseline and 7 weeks
Population: Intent-to-treat (ITT). ITT population defined as all subjects who took at least one dose of drug and had at least one ADHD-RS-IV total score available.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Vyvanse
Number analyzed (Participants) | 316
Units on a scale | -28.6 (0.61)
Statistical Analysis 1: Comparison: Vyvanse; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided

3. Secondary Outcome: Number of Participants With Improvement on Clinical Global Impression-Improvement (CGI-I)
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 or 2 on the scale.
Time Frame: 7 weeks
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Vyvanse
Number analyzed (Participants) | 316
Participants | 284

4. Secondary Outcome: Number of Participants With Improvement onParent Global Assessment (PGA)
Description: Parent Global Assessment (PGA) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: 7 weeks
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Vyvanse
Number analyzed (Participants) | 316
Participants | 267

5. Secondary Outcome: Change From Baseline in Expression and Emotional Scale for Children (EESC) Scores at 7 Weeks
Description: Expression and Emotional Scale for Children (EESC) consists of 29 items rated on a scale from 1 (not true at all) to 5 (very much true). Lower scores reflect better emotional outcomes.
Time Frame: Baseline and 7 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vyvanse
Number analyzed (Participants) | 316
Units on a scale | -7.4 (18.3)
Statistical Analysis 1: Comparison: Vyvanse; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided

6. Secondary Outcome: Changes From Baseline in Behavior Rating Inventory of Executive Function (BRIEF) Scores at 7 Weeks
Description: Behavior Rating Inventory of Executive Function (BRIEF) is an 86-item questionnaire composed of three scales (Global Executive Composite, Behavioral Recognition Index, and Metacognition Index). Items are rated 1 (never), 2 (sometimes), and 3 (often). Lower scores reflect better functioning.
Time Frame: Baseline and 7 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vyvanse
Number analyzed (Participants) | 316
Units on a scale
  Global Executive Composite | -17.9 (12.5)
  Behavioral Recognition Index | -15.4 (12.6)
  Metacognition Index | -17.6 (12.3)
Statistical Analysis 1: Comparison: Vyvanse; Global Executive Composite; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided
Statistical Analysis 2: Comparison: Vyvanse; Behavioral Recognition Index; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided
Statistical Analysis 3: Comparison: Vyvanse; Metacognition Index; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided

ADVERSE EVENTS:
Arm/Group | Vyvanse
Serious Adverse Events (participants affected / at risk) | 2/317
Other Adverse Events (participants affected / at risk) | 269/317
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vyvanse (N=317)
Syncope (Cardiac disorders) | 1 (1)
Sinus arrest (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vyvanse (N=317)
Abdominal pain upper (Gastrointestinal disorders) | 42
Nausea (Gastrointestinal disorders) | 17
Vomiting (Gastrointestinal disorders) | 17
Irritability (General disorders) | 51
Weight decreased (Investigations) | 54
Decreased appetite (Metabolism and nutrition disorders) | 137
Headache (Nervous system disorders) | 44
Affect liability (Psychiatric disorders) | 23
Initial insomnia (Nervous system disorders) | 36
Insomnia (Nervous system disorders) | 51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.